CLINICAL TRIAL: NCT06152991
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Prospective Comparative, Investigator-initiated Clinical Trial to Evaluate the Efficacy of Carnitine Orotate Complex _Godex® in Patients With Nonalcoholic Fatty Liver Disease
Brief Title: Clinical Trial Assessing Godex Carnitine Orotate Complex in Nonalcoholic Fatty Liver Disease Patients for Efficacy
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Yoon Jun Kim (Other)
Collaborators: Celltrion Pharm, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Yoon Jun Kim, Coordinating Investigator, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMTGODEX_001
Record Dates: First submitted 2023-09-21; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD; Non-Alcoholic Fatty Liver Diease; GODEX
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Double-Blindle
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This clinical trial will be conducted as a double-blind study. The double-blind condition ensures that the investigational drug and the placebo are manufactured to be indistinguishable in terms of appearance, with identical formulations and characteristics, and are supplied in identical packaging. All investigational drugs for the clinical trial will be managed using unique code numbers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Oral administration of 2 capsules of Godex® three times a day (tid) for 96 weeks
  Interventions: Drug: GODEX
- Control Group (Placebo Comparator): Oral administration of 2 placebo capsules three times a day (tid) for 96 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GODEX — The amount of active ingredient per dose (1 capsule)
  * Carnitine Orotate 150mg
  * liver extract antitoxic fraction 12.5㎎
  * Adenine Hydrochloride 2.5mg
  * Pyridoxine Hydrochloride 25mg
  * Riboflavin 0.5mg
  * Cyanocobalamin 0.125mg
  * Biphenyl Dimethyl Dicarboxylate 25mg
  Arms: Test Group
Drug: Placebo — * Anhydrous lactose 50mg.
  * Colloidal silicon dioxide 12mg.
  * Amorphous cellulose 50mg.
  * Lactose monohydrate 215.625mg.
  * Magnesium stearate 7mg.
  * Upper and lower brown opaque capsules 77mg.
  Arms: Control Group

SUMMARY:
the purpose of this clinical trial is to assess the efficacy and safety of Orotic Acid Carnitine Complex Capsules (Godex®) in comparison to a placebo control group in patients with Non-Alcoholic Fatty Liver Disease (NAFLD).

DETAILED DESCRIPTION:
the purpose of this clinical trial is to assess the efficacy and safety of Orotic Acid Carnitine Complex Capsules (Godex®) in comparison to a placebo control group in patients with Non-Alcoholic Fatty Liver Disease (NAFLD).

Godex® is being investigated for its potential to contribute to a reduction in liver fat content and improvement in liver fibrosis when administered over an extended period in patients with NAFLD. Additionally, this study aims to confirm the normalization of HbA1c and ALT, as observed in previous research, and to verify the reduction in intrahepatic fat content through MRI-PDFF analysis and improvement in liver fibrosis via MRE assessment. This investigation is motivated by the insufficient preliminary research on the long-term prescription of Godex® for NAFLD.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 to under 75, both male and female.
2. Patients with elevated liver enzymes (AST or ALT ≥ 60 or sustained AST or ALT ≥ 40 to 59 for 3 months or more).
3. For diabetic patients, those with an HbA1c level of less than 8.5% and no changes in the type and dosage of antidiabetic medications in the past 12 weeks.
4. Patients with an MRI-PDFF ≥ 7% indicating evidence of intrahepatic fat deposition, suspected of having non-alcoholic fatty liver disease.
5. Patients who voluntarily consent to participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

1. Individuals who have experienced a weight fluctuation of over 10% of their prior weight within the past 6 months.
2. Those with AST or ALT levels exceeding 10 times the upper normal limit.
3. Individuals actively involved in dieting or undergoing intense exercise therapy for weight management purposes.
4. Participants with a history of surgical weight loss procedures (e.g., bariatric surgery) or those scheduled for medical or surgical interventions for weight loss during the study period.
5. Individuals with endocrine disorders that may affect body weight (e.g., hypothyroidism, Cushing's syndrome) or those with TSH levels below 0.1uU/ml or above 10.0uU/ml in screening tests.
6. Individuals presenting evidence of chronic hepatitis, including B or C hepatitis (For B or C hepatitis, individuals with positive HBsAg or positive HCV Ab in screening tests and positive HCV RNA are included).
7. Those with a history of alcohol consumption exceeding 210 grams per week for males or 140 grams per week for females within the past year.
8. Individuals who have undergone liver transplantation.
9. Those undergoing renal dialysis or with creatinine levels exceeding twice the upper limit of normal.
10. Individuals in a medically unstable condition to the extent that they cannot participate in the clinical trial based on physical examinations across various organ systems, encompassing cardiovascular, respiratory, gastrointestinal, hepatic-biliary, metabolic, endocrine, renal-urinary, nervous, psychiatric, and other systems.
11. Individuals diagnosed with and treated for malignant tumors within the past 5 years (excluding basal cell carcinoma or squamous cell carcinoma of the skin, provided it has been determined as "cured" after surgery or treatment at the investigator's discretion).
12. Pregnant or lactating women or fertile women who do not consent to using effective contraceptive methods during the study period (oral contraceptives are not considered an effective contraceptive method).
13. Patients currently receiving levodopa.
14. Individuals with genetic conditions such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
15. Individuals with a history of significant alcohol or substance misuse within the past year.
16. hose who have taken medications containing UDCA (Ursodeoxycholic acid), dimethyl-4,4'-dimethoxy-5,6,5',6'-dimethendixoybiphenyl-2,2'-dicarboxylate (DDB), or silymarin components within 4 weeks before the first dose.
17. Those who have taken vitamin E (≥ 800 IU/day), received pioglitazone therapy, or used drugs approved for NASH treatment within 12 weeks before the first dose (exceptions granted if a stable dosage has been maintained for the past 24 weeks).
18. Those who have taken medications affecting body weight within 12 weeks before the first dose, including obesity treatments (absorption inhibitors and appetite suppressants), antidepressants, contraceptives, oral steroids, amphetamines, phentermine, sibutramine, female hormones, thyroid hormones, etc. (exceptions granted if a stable dosage has been maintained for the past 24 weeks).
19. Other individuals deemed unsuitable by the Principal Investigator
20. Those who have taken investigational drugs for other clinical trials within the last 6 months.

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Change in intrahepatic fat content measured by MRI-PDFF | 48-week time point compared to baseline.
  For each group, the mean and standard deviation [if necessary, median and interquartile range (IQR)] along with a 95% confidence interval are provided for the liver fat content measured by MRI-PDFF at baseline and the change from baseline to the 48-week time point. The difference in liver fat content at baseline and the change in liver fat content at the 48-week time point between the two groups are tested using the two-sample t-test or Wilcoxon's rank sum test, depending on the normality of the data.

SECONDARY OUTCOMES:
Changes in hepatic fibrosis measured by MRE at 96 weeks compared to baseline. | 96-week time point compared to baseline.
  Present the mean and standard deviation [or median and IQR (Inter Quartile Range), if necessary] along with a 95% confidence interval for the intrahepatic fat measured by MRI-PDFF at baseline and the change from baseline to week 48 for each group. The comparison of intrahepatic fat at baseline and the change in intrahepatic fat at week 48 between the two groups will be assessed using two sample t-test or Wilcoxon's rank sum test, depending on the normality of the data.
Changes in hepatic fat content measured by MRI-PDFF at 96 weeks compared to baseline. | 96-week time point compared to baseline.
  Present the mean and standard deviation (or median and IQR, if necessary) along with a 95% confidence interval for the intrahepatic fat measured by MRI-PDFF at baseline and at week 96, as well as the change from baseline to week 96 for each group. The comparison of intrahepatic fat at baseline and the change in intrahepatic fat at week 96 between the two groups will be assessed using two-sample t-test or Wilcoxon's rank-sum test, depending on the normality of the data.
Proportion of subjects with a reduction in hepatic fat content measured by MRI-PDFF at 48 and 96 weeks of 20% or more compared to baseline. | 96-week time point compared to baseline.
  * The percentage of subjects with a reduction of 20% or more in intrahepatic fat, as measured by MRI-PDFF at baseline compared to weeks 48 and 96, will be defined based on the % change. If the % change is 20% or greater, it will be considered a reduction.
  * The comparison between the trial group and the control group regarding the percentage of subjects with a reduction of 20% or more in intrahepatic fat, as measured by MRI-PDFF at baseline compared to weeks 48 and 96, will be analyzed using Pearson's chi-square test or Fisher's exact test.
  * Additionally, the reduction in intrahepatic fat will be categorized into three intervals: less than 20%, 30-50%, and 50% or more. The percentage of subjects with reduced intrahepatic fat in each interval for both the trial group and the control group will be compared using Pearson's chi-square test or Fisher's exact test.t.
Proportion of subjects with an improvement in hepatic fibrosis measured by MRE at 96 weeks of 20% or more compared to baseline. | 48-week and 96-week time points compared to baseline.
  * The percentage of subjects showing an improvement in liver fibrosis of 20% or more, as measured by MRE at baseline compared to week 96, will be defined based on the % change. An improvement will be considered when the % change is -20% or less.
  * A comparative analysis between the test group and the control group regarding the percentage of subjects with an improvement in liver fibrosis of 20% or more, as measured by MRE at baseline compared to week 96, will be conducted using either Pearson's chi-square test or Fisher's exact test.
Changes in CAP measured by Fibroscan at 48 and 96 weeks compared to baseline. | 96-week time point compared to baseline.
  The mean and 95% confidence intervals for the changes in CAP (Controlled Attenuation Parameter) measured by Fibroscan at baseline compared to week 48 and week 96 are presented. Data normality will be assessed, and either a two-sample t-test or Wilcoxon's rank-sum test will be employed to perform a comparative analysis of the changes in CAP measured by Fibroscan at baseline compared to week 48 and week 96 between the test group and the control group.
Changes in LSM measured by Fibroscan at 48 and 96 weeks compared to baseline. | 96-week time point compared to baseline.
  The mean and 95% confidence intervals for the changes in LSM (Liver Stiffness Measurement) measured by Fibroscan at baseline compared to week 48 and week 96 are presented. Data normality will be assessed, and either a two-sample t-test or Wilcoxon's rank-sum test will be employed to perform a comparative analysis of the changes in LSM measured by Fibroscan at baseline compared to week 48 and week 96 between the test group and the control group.
Changes in body weight at 48 and 96 weeks compared to baseline. | 48-week and 96-week time points compared to baseline.
  Mean and 95% confidence intervals for changes in body weight at baseline compared to weeks 48 and 96 are provided. Data normality will be assessed, and either a two-sample t-test or Wilcoxon's rank-sum test will be used to perform a comparative analysis of changes in body weight at baseline compared to weeks 48 and 96 between the test group and the control group.
Changes in waist circumference at 48 and 96 weeks compared to baseline. | 48-week and 96-week time points compared to baseline.
  Mean and 95% confidence intervals for changes in body waist circumference at baseline compared to weeks 48 and 96 are provided. Data normality will be assessed, and either a two-sample t-test or Wilcoxon's rank-sum test will be used to perform a comparative analysis of changes in waist circumference at baseline compared to weeks 48 and 96 between the test group and the control group.
Changes in AST, ALT, r-GTP, and normalization rates at 48 and 96 weeks compared to baseline. | 48-week and 96-week time points compared to baseline.
  * Mean and 95% confidence intervals for changes in AST, ALT, and r-GTP at baseline compared to weeks 48 and 96 are provided. Data normality will be assessed, and either a two-sample t-test or Wilcoxon's rank-sum test will be used to perform a comparative analysis of changes in AST, ALT, and r-GTP at baseline compared to weeks 48 and 96 between the test group and the control group.
  * The proportion of subjects in the test group and the control group with normalization of AST, ALT, and r-GTP at weeks 48 and 96 will be compared using Pearson's chi-square test or Fisher's exact test.
Changes in HOMA-IR ≥2.0 at 48 and 96 weeks compared to baseline | 48-week and 96-week time points compared to baseline.
  - Mean and 95% confidence intervals for changes in insulin resistance (insulin resistance HOMA-IR ≥2.0) at baseline compared to weeks 48 and 96 are provided. Data normality will be assessed, and either a two-sample t-test or Wilcoxon's rank-sum test will be used to perform a comparative analysis of changes in insulin resistance (insulin resistance HOMA-IR ≥2.0) at baseline compared to weeks 48 and 96 between the test group and the control group.
Changes in glycated hemoglobin (HbA1c) at 48 and 96 weeks compared to baseline | 48-week and 96-week time points compared to baseline.
  - Mean and 95% confidence intervals for changes in glycated hemoglobin (HbA1c) at baseline compared to weeks 48 and 96 are provided. Data normality will be assessed, and either a two-sample t-test or Wilcoxon's rank-sum test will be used to perform a comparative analysis of changes in glycated hemoglobin, at baseline compared to weeks 48 and 96 between the test group and the control group.
Changes in fasting blood glucose at 48 and 96 weeks compared to baseline | 48-week and 96-week time points compared to baseline.
  - Mean and 95% confidence intervals for changes in fasting blood glucose at baseline compared to weeks 48 and 96 are provided. Data normality will be assessed, and either a two-sample t-test or Wilcoxon's rank-sum test will be used to perform a comparative analysis of changes in fasting blood glucose at baseline compared to weeks 48 and 96 between the test group and the control group.
Changes in lipid profiles (total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides) at 48 and 96 weeks compared to baseline. | 48-week and 96-week time points compared to baseline.
  - Mean and 95% confidence intervals for changes in lipid profiles at baseline compared to weeks 48 and 96 are provided. Data normality will be assessed, and either a two-sample t-test or Wilcoxon's rank-sum test will be used to perform a comparative analysis of changes in lipid profiles at baseline compared to weeks 48 and 96 between the test group and the control group.
Incidence of NAFLD risk factor diseases (hypertension, diabetes, dyslipidemia, etc.) at 48 and 96 weeks compared to baseline. | 48-week and 96-week time points compared to baseline.
  - Frequencies and incidence rates of NAFLD risk factor-related diseases in the test group and control group at baseline compared to weeks 48 and 96 are calculated, and 95% confidence intervals are provided. Pearson's chi-square test or Fisher's exact test will be used to analyze the difference in the incidence rates of NAFLD risk factor-related diseases at weeks 48 and 96 between the test group and the control group.
Rate of medication discontinuation due to adverse events. | during the intervention
  - The frequency and proportion of subjects who discontinued medication due to adverse events are presented according to adverse cases. The difference in medication discontinuation rates due to adverse events between the two groups will be compared using Pearson's chi-square test or Fisher's exact test.

OTHER OUTCOMES:
Adverse events | immediately after the intervention
  - The summary and analysis of adverse events are conducted for treatment-emergent adverse events (TEAEs) occurring after the administration of investigational medicinal products in the clinical trial. The frequency and percentage of adverse events, adverse drug reactions (ADRs), and serious adverse events (SAEs) occurring after the administration of investigational medicinal products are presented by treatment group. These occurrences are compared using Pearson's chi-square test or Fisher's exact test
Proportion of subjects with abnormal Laboratory Tests | immediately after the intervention
  - Within-group and between-group comparisons are conducted. For within-group comparisons between the test group and the control group, continuous variables are analyzed using paired t-tests or Wilcoxon's signed-rank test depending on whether the normality assumption is satisfied, and categorical variables are analyzed using McNemar's test. For between-group comparisons between the test group and the control group, continuous variables are analyzed based on the normality assumption by confirming the normality of the data and using either the two-sample t-test or Wilcoxon's rank sum test, while categorical variables are analyzed using Pearson's chi-square test or Fisher's exact test.
Proportion of subjects with abnormal vital signs | immediately after the intervention
  - Within-group and between-group comparisons are conducted. For within-group comparisons between the test group and the control group, continuous variables are analyzed using paired t-tests or Wilcoxon's signed-rank test depending on whether the normality assumption is satisfied, and categorical variables are analyzed using McNemar's test. For between-group comparisons between the test group and the control group, continuous variables are analyzed based on the normality assumption by confirming the normality of the data and using either the two-sample t-test or Wilcoxon's rank sum test, while categorical variables are analyzed using Pearson's chi-square test or Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: YoonJun Kim, MD.PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea